CLINICAL TRIAL: NCT02355743
Title: Prophylactic Recombinant Tissue Plasminogen Activator in the Prevention of Central Venous Access Device (CVAD)-Associated Thrombosis and Infection in Pediatric Patients With Short Bowel Syndrome
Brief Title: rtPA in in the Prevention of CVAD-Associated Thrombosis and Infection in Pediatric Patients With Short Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lynn Malec (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Lynn Malec, Assistant Professor of Medicine and Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO13120030
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rtPA lock therapy Recipients (Experimental): rtPA 2 mg/2 ml, or 110% of the volume of the catheter lumen if less than 2 mL, administered locally in a volume to fill the lumen (dead space) of the CVAD, once weekly for a total of 24 weeks
  Interventions: Drug: rtPA lock therapy

INTERVENTIONS:
Drug: rtPA lock therapy — rtPA 2 mg/2 ml, or 110% of the volume of the catheter lumen if less than 2 mL, administered locally in a volume to fill the lumen (dead space) of the CVAD, once weekly for a total of 24 weeks. rtPA will be given as research intervention as "lock therapy" in that it will dwell within the catheter of the CVAD for a specified duration of time and then be removed (aspirated); in this setting the medication is not given to the patient as a flush, i.e. in systemic fashion.
  Other Names: rtPA

SUMMARY:
The primary research question is, in patients with short bowel syndrome requiring central venous access device (CVAD) for long-term total parenteral nutrition, is once weekly recombinant tissue plasminogen activator (rtPA) lock therapy more effective than routine care using heparin flushes in reducing the incidence of line-associated thrombosis and infection.

DETAILED DESCRIPTION:
Central venous access devices (CVAD) are used routinely in chronically ill pediatric patients for administration of medications, parenteral nutrition and laboratory testing. Several complications resulting from the use of long-term CVADs, namely venous sepsis and thrombosis, can significantly increase associated morbidity and mortality. CVAD-associated thrombosis occurs in up to 50% of children with long-term CVAD use and this is especially common in patients requiring life-sustaining long-term total parenteral nutrition (1). Catheter thrombosis may arise from fibrin sheath formation around the catheter tip, intraluminal blood clot within the catheter, or venous thrombosis obstructing the vein and occluding the catheter tip. Within 24 hours and typically within 2 weeks of placement of a CVAD, a fibrin sheath forms around its tip (2-5). Development of intraluminal thrombosis or venous thrombosis is less predictable.

There is a growing body of evidence linking the development of CVAD-associated thrombosis and line-related infection. It is known that proteins within the thrombus including fibronectin and fibrinogen attract bacteria, specifically staphylococcal species. The bacteria bind to ligands associated with the thrombus thus allowing for bacterial proliferation (6-8). The clinical relevance of line thrombus in development of line infection is underscored in a study of pediatric patients with Hickman catheters, of whom 18% with catheter thrombosis developed a line-associated bloodstream infection, while none developed a catheter infection that did not also have a catheter clot (7). Thus, we hypothesize that prevention of catheter-related clot formation with use of a local thrombolytic agent will also prevent infection in the catheter.

The primary research question we pose is, in patients with short bowel syndrome requiring central venous access device (CVAD) for long-term total parenteral nutrition, is once weekly recombinant tissue plasminogen activator (rtPA) lock therapy more effective than routine care using heparin flushes in reducing the incidence of line-associated thrombosis and infection.

ELIGIBILITY:
Inclusion Criteria:

1. subjects with short bowel syndrome
2. requirement for central venous access device (CVAD) for long-term TPN administration
3. age >/= 6 months to < 16 years
4. ability to initiate rtPA during hospitalization for newly inserted CVAD
5. ability to be enrolled within 48 hours of CVAD placement.

Exclusion Criteria:

1. platelet count <50,000
2. active bleeding
3. age =/> 16 years at time of consent.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2016-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Malec, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Children's Hospital of Pittsburgh of UPMC inpatient setting
Pre-assignment Details: All patients received study intervention of rtPA lock therapy which was initiated within 48 hours of a new central venous access device being placed.
Period: Overall Study
Arm/Group | rtPA Lock Therapy Recipients
Started | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | rtPA Lock Therapy Recipients
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 4.4 [1.4 to 11.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Central venous access device associated infections in prior 6 months [Median (Inter-Quartile Range); unit: infections] | 2 [0.8 to 2.5]
Hospitalizations in prior 6 months [Mean (Inter-Quartile Range); unit: hospitalizations] | 3 [1.8 to 4.5]
Lifetime number of central venous access devices [Median (Inter-Quartile Range); unit: central venous access devices] | 6.5 [3 to 14]
Central venous access devices in prior 6 months [Median (Inter-Quartile Range); unit: central venous access devices] | 2 [1.8 to 3.3]

OUTCOME MEASURES:

1. Primary Outcome: Development of CVAD Line Thrombosis
Description: This will be defined as a thrombosis that is discovered due to clinical findings concerning for a possible thrombosis as identified by the treating physician including, but not limited to, swelling, color change, or pain in the extremity, CVAD not providing blood return and/or being able to be flushed.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: thromboses
Arm/Group | rtPA Lock Therapy Recipients
Number analyzed (Participants) | 6
thromboses | 0 [0 to 0]

2. Secondary Outcome: Development of Line-associated Infection
Description: This will be defined as a line associated infection not related to other co-infection (i.e. such as pneumonia, UTI)
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: infections
Arm/Group | rtPA Lock Therapy Recipients
Number analyzed (Participants) | 6
infections | 0.5 [0 to 1]

3. Secondary Outcome: Need for Central Line Replacement
Description: This will be defined as a line removal and replacement due to infection, malfunction or other issues
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: line replacements
Arm/Group | rtPA Lock Therapy Recipients
Number analyzed (Participants) | 6
line replacements | 1 [0 to 2.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a course of 6 months
Arm/Group | rtPA Lock Therapy Recipients
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No